CLINICAL TRIAL: NCT01176565
Title: Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH)-II: A Phase III Randomized Multicenter Clinical Trial of Blood Pressure Reduction for Hypertension in Acute Intracerebral Hemorrhage
Brief Title: Antihypertensive Treatment of Acute Cerebral Hemorrhage-II
Acronym: ATACH-II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Planned interim analysis: no significant outcome differences between groups
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medical University of South Carolina (Other); Johns Hopkins University (Other); University of Michigan (Other); Neurocritical Care Research Network (Unknown); National Cerebral and Cardiovascular Center, Japan (Other); Japan Cardiovascular Research Foundation (Other); Beijing Tiantan Hospital (Other); China Medical University Hospital (Other); University Hospital Heidelberg (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1207M17921; U01NS062091 (NIH); U01NS061861 (NIH); U01NS059041 (NIH); U01NS056975 (NIH); H23-4-3 (Other Grant/Funding Number: Intramural Research Fund for Cardiovascular Diseases of the National Cerebral and Cardiovascular Center, Japan)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: Acute hypertensive response; intracerebral hemorrhage; blood pressure; outcome; nicardipine
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Nicardipine

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomized 1:1 via computer-generated treatment assignment within 4.5 hours of neurological symptom onset to either standard or intensive SBP management using intravenous nicardipine hydrochloride as the primary BP control agent through 24 hours from randomization. Enrolled patients from both treatment arms are otherwise treated similarly after 24 hours, according to their medical needs. Standards of care management for spontaneous intracerebral hemorrhage published in the 2010 American Heart Association guidelines are incorporated in to the study protocol. All enrolled patients are followed through 90 days (± 14 days per protocol window; up to ± 30 days data is used) unless death or withdrawal occurs sooner. Primary analysis based on intent-to-treat (ITT) principles.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The trial intervention is conducted open-label to avoid concealing clinically necessary patient blood pressure and intravenous drug administration information. Clinical data including SBP values are primarily taken from entries recorded in to the patient's official medical record by hospital staff and are independently monitor-verified. Assessors for the primary outcome (mRS) at 90 days are are unaware of the treatment assignment or in-hospital clinical course of the subjects assessed. De-identified imaging studies are coded independently of subject number so the central imaging reader is unaware of the treatment assignment, clinical findings, or time points of image acquisition for data recorded from imaging. The study (lead) principal investigator and leadership committee members are unable to associate the treatment assignment of subjects to their outcomes or adverse events for purposes of trial decision-making. Adverse events are adjudicated by an independent oversight committee.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard SBP Reduction Arm (Active Comparator): Intravenous nicardipine hydrochloride will be used as necessary (pro re nata or "PRN") as the primary agent in lowering SBP.
  The goal for the standard BP reduction group will be to reduce and maintain SBP < 180 mmHg for 24 hours from randomization. 160 mmHg is the target SBP for this arm.
  For the standard group, SBP below the assigned treatment range is not artificially elevated to stay within the range if lower SBP occurs with nicardipine turned off (no fluid bolus given unless SBP falls below 110 mmHg with nicardipine off and there is risk for hypotension). Euvolemic fluid maintenance is encouraged for all patients according to their medical needs, which may differ.
  Interventions: Drug: Intravenous nicardipine hydrochloride
- Intensive SBP Reduction Arm (Active Comparator): Intravenous nicardipine hydrochloride will be used as necessary (pro re nata or "PRN") as the primary agent in lowering SBP.
  The goal for the intensive BP reduction group will be to reduce and maintain SBP < 140 mmHg for 24 hours from randomization. 125 mmHg is the target SBP for this arm.
  For the intensive group, SBP falling below 110 mmHg (lower limit of the assigned treatment range) with nicardipine off is treated with normal saline fluid bolus to prevent or remedy hypotension. Euvolemic fluid maintenance is encouraged for all patients according to their medical needs, which may differ.
  Interventions: Drug: Intravenous nicardipine hydrochloride

INTERVENTIONS:
Drug: Intravenous nicardipine hydrochloride — IV nicardipine is initiated at a rate of 5 mg/hr, is continued, and is increased by 2.5 mg/hr increments every 15 min until the target SBP or maximum dose of 15 mg/hr is reached. If SBP is above the target SBP despite infusion of the maximum nicardipine dose for 30 minutes, a second agent may be used (Labetalol 5-20 mg IV bolus every 15 min; diltiazem/urapidil in countries without labetalol) for another hour. Nicardipine infusion is decreased incrementally or is stopped if SBP falls below the desired treatment range.
  Fluid bolus for SBP still falling below 110 mmHG (millimeters of mercury) with nicardipine off is given to prevent organ hypoperfusion. Vasopressor agents are not used unless symptoms related to or possibly exacerbated by hypoperfusion are present.
  Other Names: Cardene® I.V.; Nicardipine HCl injection; nicardipine hydrochloride injection; nicardipine IV; nicardipine; nicardipine hydrochloride

SUMMARY:
The specific aims of this study are to:

1. Definitively determine the therapeutic benefit of the intensive treatment relative to the standard treatment in the proportion of patients with death and disability (mRS 4-6) at 3 months among subjects with ICH who are treated within 4.5 hours of symptom onset.
2. Evaluate the therapeutic benefit of the intensive treatment relative to the standard treatment in the subjects' quality of life as measured by EuroQol at 3 months.
3. Evaluate the therapeutic benefit of the intensive treatment relative to the standard treatment in the proportion of hematoma expansion (defined as increase from baseline hematoma volume of at least 33%) and in the change from baseline peri-hematoma volume at 24 hours on the serial computed tomographic (CT) scans.
4. Assess the safety of the intensive treatment relative to the standard treatment in the proportion of subjects with treatment-related serious adverse events (SAEs) within 72 hours.

DETAILED DESCRIPTION:
The report from a National Institute of Neurological Disorders and Stroke Workshop on priorities for clinical research in intracerebral hemorrhage (ICH) in December 2003 recommended clinical trials for evaluation of blood pressure (BP) management in acute ICH as a leading priority. The Special Writing Group of the Stroke Council of the American Heart Association in 1999 and 2007 emphasized the need for clinical trials to ensure evidence-based treatment of acute hypertension in ICH. Consequently, we propose to conduct a five-year international, multicenter, open-labeled, randomized, controlled, Phase III trial to determine the efficacy of early, intensive antihypertensive treatment using intravenous nicardipine for acute hypertension in subjects with co-morbid hypertension and spontaneous supratentorial ICH. The primary hypothesis of this large, streamlined, focused trial is that the group treated with intensive BP reduction (systolic BP [SBP] of 140 mmHg or less - hereafter referred to as the intensive treatment) using intravenous nicardipine infusion for 24 hours reduces the proportion of death and disability at 3 months by 10% or greater compared with the group treated with the standard BP reduction (SBP of 180 mmHg or less - hereafter referred to as the standard treatment) among patients with ICH treated within 4.5 hours of symptom onset. The underlying mechanism for this expected beneficial effect of intensive treatment is mediated through reduction of the rate and magnitude of hematoma expansion observed in approximately 38% of patients with acute ICH. The trial will recruit a maximum of 1,280 subjects with ICH who meet the eligibility criteria. The primary outcome is the proportion of death and disability at 3 months defined by modified Rankin scale (mRS) score of 4 to 6. The proposed clinical trial is the natural extension of numerous case series, a subsequent pilot trial funded by the National Institutes of Health National Institute of Health (NIH), and a preliminary randomized controlled trial in this patient group funded by the Australian National Health and Medical Research Council, that have recently confirmed the safety and tolerability of both the regimen and goals of the antihypertensive treatment in acutely hypertensive patients with ICH proposed in the present trial. The proposed trial will have important public health implications by providing necessary information regarding the efficacy and safety of antihypertensive treatment of acute hypertension observed in up to 75% of the subjects with ICH. BP treatment represents a strategy that can be made widely available without the need of specialized equipment and personnel and therefore can make a major impact upon outcome in patients with ICH. Substantial reduction in morbidity and mortality appears possible if the estimates of treatment effect sizes from current pilot trials are accurate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* IV nicardipine can be initiated within 4.5 hours of symptom onset.
* Clinical signs consistent with the diagnosis of stroke, including impairment of language, motor function, cognition, and/or gaze, vision, or neglect.
* Total Glasgow Coma Scale (GCS) score (aggregate of verbal, eye, and motor response scores) of 5 or greater at time of emergency department (ED) arrival.
* International normalized ratio (INR) value < 1.5
* CT scan demonstrates intraparenchymal hematoma with manual hematoma volume measurement <60 cc.
* For subjects randomized prior to IV antihypertensive administration: SBP greater than 180 mmHg* prior to IV antihypertensive treatment (this includes pre-hospital treatment) AND WITHOUT spontaneous SBP reduction to below 180 mmHg at the time of randomization OR
* For subjects randomized after IV antihypertensive administration: SBP greater than 180 mmHg* prior to IV antihypertensive treatment (this includes pre-hospital treatment) AND WITHOUT SBP reduction to below 140 mmHg at the time of randomization.
* Informed consent obtained by subject, legally authorized representative, or next of kin.

  * Notes: The unit "mmHg" stands for "millimeters of mercury", a standard way of measuring blood pressure. Patients with SBP < 180 mmHg should be monitored for 4.5 hours from symptom onset as their SBP may rise to eligible levels before the eligibility window closes.

Exclusion Criteria:

* ICH is due to previously known neoplasms, arteriovenous malformation (AVM), or aneurysms.
* Intracerebral hematoma considered to be related to trauma.
* ICH located in infratentorial regions such as pons or cerebellum.
* Intraventricular hemorrhage (IVH) associated with intraparenchymal hemorrhage and blood completely fills one lateral ventricle or more than half of both ventricles.
* Patient to receive immediate surgical evacuation.
* Current pregnancy, or parturition within previous 30 days, or active lactation.
* Use of dabigatran within the last 48 hours**.
* A platelet count less than 50,000 per microliter (µL or mm3)
* Known sensitivity to nicardipine.
* Pre-morbid disability requiring assistance in ambulation or activities of daily living.
* Subject's living will precludes aggressive ICU management.
* Subject is currently participating in another interventional clinical trial

  * Use of dabigatran was clarified through investigator presentations, educational materials, and clinical tools to include newer similar class medications (such as rivaroxaban, apixaban, and edoxaban) that were being developed and in various stages of approval across enrolling countries through the course of this trial, in the event that patients using these medications may have been encountered during screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-05-15 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2016-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan I Qureshi, MD, Study Chair — University of Minnesota; Yuko Y Palesch, PhD, Study Director — Medical University of South Carolina; Adnan I Qureshi, MD, Principal Investigator — University of Minnesota; Yuko Y Palesch, PhD, Principal Investigator — Medical University of South Carolina
Locations (171):
- United States (116):
  - UAB Comprehensive Stroke Center, Birmingham, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - Mayo Clinic Pheonix, Scottsdale, Arizona
  - Banner University Medical Center - South Campus, Tuscon, Arizona
  - Banner University Medical Center - University Campus, Tuscon, Arizona
  - Community Regional Medical Center of Fresno, Fresno, California
  - University of California San Diego, La Jolla, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Good Samaritan Hospital, San Jose, California
  - Santa Clara Valley Medical Center, Santa Clara, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - University of Florida Gainesville, Gainesville, Florida
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Eastern Idaho Medical Consultants, Idaho Falls, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Southern Illinois University Memorial Medical Center, Springfield, Illinois
  - Lutheran Hospital Indiana, Fort Wayne, Indiana
  - Parkview Hospital, Fort Wayne, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - West Jefferson Medical Center, Marrero, Louisiana
  - Interim LSU Hospital, New Orleans, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Shreveport, Louisiana
  - Maine Medical Center, South Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Wayne State University - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Essentia Health St. Mary's Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Neuroscience Institute, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - St. Joseph's Regional Medical Center, Clifton, New Jersey
  - New Jersey Neuroscience Institute, JFK Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - New York City Health and Hospitals Corp. / Kings County Hospital, Brooklyn, New York
  - Mamoides Medical Center, Brooklyn, New York
  - Sister of Charity/Buffalo Mercy Hospital, Catholic Health System, Buffalo, New York
  - UHS Wilson Medical Center, Johnson City, New York
  - North Shore University Hospital, Manhasset, New York
  - SUNY Downstate, New York, New York
  - Columbia University, New York, New York
  - Lincoln Medical and Mental Health Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Strong Stroke Center, Rochester, New York
  - Mission Hospital, Asheville, North Carolina
  - Guilford Neurologic Associates, Greenboro, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Novant Clinical Research Institute/Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center (Wake Forest School of Medicine), Winston-Salem, North Carolina
  - Akron General Hospital, Akron, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University - Wexner Medical Center, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oklahoma University Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - Providence Brain and Spine Institute, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Univ/ Hershey Med Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wellspan York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health, Columbia, South Carolina
  - Vanderbilt Stroke Center, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - St. David's Medical Center, Austin, Texas
  - University Medical Center Brackenridge, Austin, Texas
  - UT Southwestern - Parkland Hospital, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - Memorial Herman - Texas Medical Center, Houston, Texas
  - Baylor College of Medicine - Ben Taub Community Hospital, Houston, Texas
  - Baylor College of Medicine - St. Luke's Episcopal Hospital, Houston, Texas
  - Methodist Hospital - The Neurological Institute, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - West Virginia University - Ruby Memorial Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwakee, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- China (12):
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Baotou Central Hospital, Baotou
  - Beijing Tiantan Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Datong Third People's Hospital, Datong
  - The First Hospital of Shanxi Medical University, Taiyuan
  - The First People's Hospital of Taizhou, Taizhou
  - Tianjin Fourth Central Hospital, Tianjin
  - Wuhan Brain Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - People's Hopital of Zhengzhou, Zhengzhou
- Germany (10):
  - Charité Universtity Medicine Berlin, Berlin
  - University of Bonn, Bonn
  - University Hospital Dresden, Dresden
  - Clinic Frankfurt Hoechst, Frankfurt
  - University Hospital Halle, Halle
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Leipzig, Leipzig
  - University Hospital Mannheim, Mannheim
  - University Hospital Meunster, Münster
  - University of Tubingen, Tübingen
- Japan (16):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Saiseikai Yokohamashi Tobu Hospital, Kanagawa, Kanagowa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kyushu Medical Center, Fukuoka
  - Gifu University Hospital, Gifu
  - St. Marianna - Toyoko, Kawasaki
  - St. Marianna University Hospital, Kawasaki
  - Kobe City Medical Center General Hospital, Kobe
  - Kawasaki Medical School, Okayama
  - National Cerebral and Cardiovascular Center, Osaka
  - Kohnan Hospital, Sendai
  - Toranomon Hospital, Tokyo
  - Saiseikai Central Hospital - Tokyo, Tokyo
  - Keio University Hospital, Tokyo
  - Kyorin University, Tokyo
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Boramae Hospital, Seoul
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hopital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Shin-Kong Wu Ho-Su Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Veteran's Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
A public use data set from the study database will be made available. A process for sharing subject head imaging studies that may be associated with the data set is under evaluation.

REFERENCES:
- [Background] Qureshi AI, Palesch YY, Martin R, Novitzke J, Cruz-Flores S, Ehtisham A, Ezzeddine MA, Goldstein JN, Hussein HM, Suri MF, Tariq N; Antihypertensive Treatment of Acute Cerebral Hemorrhage Study Investigators. Effect of systolic blood pressure reduction on hematoma expansion, perihematomal edema, and 3-month outcome among patients with intracerebral hemorrhage: results from the antihypertensive treatment of acute cerebral hemorrhage study. Arch Neurol. 2010 May;67(5):570-6. doi: 10.1001/archneurol.2010.61. PMID 20457956
- [Background] Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH) investigators. Antihypertensive treatment of acute cerebral hemorrhage. Crit Care Med. 2010 Feb;38(2):637-48. doi: 10.1097/CCM.0b013e3181b9e1a5. PMID 19770736
- [Background] Qureshi AI. Acute hypertensive response in patients with stroke: pathophysiology and management. Circulation. 2008 Jul 8;118(2):176-87. doi: 10.1161/CIRCULATIONAHA.107.723874. No abstract available. PMID 18606927
- [Background] Qureshi AI. Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH): rationale and design. Neurocrit Care. 2007;6(1):56-66. doi: 10.1385/ncc:6:1:56. PMID 17356194
- [Background] Qureshi AI, Palesch YY. Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH) II: design, methods, and rationale. Neurocrit Care. 2011 Dec;15(3):559-76. doi: 10.1007/s12028-011-9538-3. PMID 21626077
- [Background] Qureshi AI, Palesch YY, Martin R, Novitzke J, Cruz Flores S, Ehtisham A, Goldstein JN, Kirmani JF, Hussein HM, Suri MF, Tariq N; Antihypertensive Treatment of Acute Cerebral Hemorrhage Investigators. Systolic blood pressure reduction and risk of acute renal injury in patients with intracerebral hemorrhage. Am J Med. 2012 Jul;125(7):718.e1-6. doi: 10.1016/j.amjmed.2011.09.031. Epub 2012 May 4. PMID 22560810
- [Background] Qureshi AI, Palesch YY, Martin R, Toyoda K, Yamamoto H, Wang Y, Wang Y, Hsu CY, Yoon BW, Steiner T, Butcher K, Hanley DF, Suarez JI. Interpretation and Implementation of Intensive Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial (INTERACT II). J Vasc Interv Neurol. 2014 Jun;7(2):34-40. No abstract available. PMID 25132910
- [Result] Qureshi AI, Palesch YY, Barsan WG, Hanley DF, Hsu CY, Martin RL, Moy CS, Silbergleit R, Steiner T, Suarez JI, Toyoda K, Wang Y, Yamamoto H, Yoon BW; ATACH-2 Trial Investigators and the Neurological Emergency Treatment Trials Network. Intensive Blood-Pressure Lowering in Patients with Acute Cerebral Hemorrhage. N Engl J Med. 2016 Sep 15;375(11):1033-43. doi: 10.1056/NEJMoa1603460. Epub 2016 Jun 8. PMID 27276234
- [Derived] Li Q, Lv X, Morotti A, Qureshi AI, Dowlatshahi D, Falcone GJ, Sheth KN, Shoamanesh A, Murthy SB, Viswanathan A, Goldstein JN. Optimal Magnitude of Blood Pressure Reduction and Hematoma Growth and Functional Outcomes in Intracerebral Hemorrhage. Neurology. 2025 Mar 11;104(5):e213412. doi: 10.1212/WNL.0000000000213412. Epub 2025 Feb 6. PMID 39913881
- [Derived] Tsukita K, Sakamaki-Tsukita H, Kaiser S, Zhang L, Messa M, Serrano-Fernandez P, Takahashi R. High-Throughput CSF Proteomics and Machine Learning to Identify Proteomic Signatures for Parkinson Disease Development and Progression. Neurology. 2023 Oct 3;101(14):e1434-e1447. doi: 10.1212/WNL.0000000000207725. Epub 2023 Aug 16. PMID 37586882
- [Derived] Qureshi AI, Huang W, Hanley DF, Hsu CY, Martin RH, Malhotra K, Steiner T, Suarez JI, Yamamoto H, Toyoda K. Early Hyperchloremia is Independently Associated with Death or Disability in Patients with Intracerebral Hemorrhage. Neurocrit Care. 2022 Oct;37(2):487-496. doi: 10.1007/s12028-022-01514-2. Epub 2022 May 5. PMID 35513751
- [Derived] Tanaka K, Koga M, Fukuda-Doi M, Qureshi AI, Yamamoto H, Miwa K, Ihara M, Toyoda K; ATACH-2 Trial Investigators. Temporal Trajectory of Systolic Blood Pressure and Outcomes in Acute Intracerebral Hemorrhage: ATACH-2 Trial Cohort. Stroke. 2022 Jun;53(6):1854-1862. doi: 10.1161/STROKEAHA.121.037186. Epub 2022 Apr 11. PMID 35400202
- [Derived] Tsukita K, Sakamaki-Tsukita H, Takahashi R. Long-term Effect of Regular Physical Activity and Exercise Habits in Patients With Early Parkinson Disease. Neurology. 2022 Feb 22;98(8):e859-e871. doi: 10.1212/WNL.0000000000013218. Epub 2022 Jan 12. PMID 35022304
- [Derived] Magid-Bernstein JR, Li Y, Cho SM, Piran PJ, Roh DJ, Gupta A, Shoamanesh A, Merkler A, Zhang C, Avadhani R, Montano N, Iadecola C, Falcone GJ, Sheth KN, Qureshi AI, Rosand J, Goldstein J, Awad I, Hanley DF, Kamel H, Ziai WC, Murthy SB. Cerebral Microbleeds and Acute Hematoma Characteristics in the ATACH-2 and MISTIE III Trials. Neurology. 2022 Mar 8;98(10):e1013-e1020. doi: 10.1212/WNL.0000000000013247. Epub 2021 Dec 22. PMID 34937780
- [Derived] Qureshi AI, Huang W, Lobanova I, Chandrasekaran PN, Hanley DF, Hsu CY, Martin RH, Steiner T, Suarez JI, Yamamoto H, Toyoda K. Effect of Moderate and Severe Persistent Hyperglycemia on Outcomes in Patients With Intracerebral Hemorrhage. Stroke. 2022 Apr;53(4):1226-1234. doi: 10.1161/STROKEAHA.121.034928. Epub 2021 Nov 30. PMID 34844422
- [Derived] Miwa K, Koga M, Fukuda-Doi M, Yamamoto H, Tanaka K, Yoshimura S, Ihara M, Qureshi AI, Toyoda K. Effect of Heart Rate Variabilities on Outcome After Acute Intracerebral Hemorrhage: A Post Hoc Analysis of ATACH-2. J Am Heart Assoc. 2021 Aug 17;10(16):e020364. doi: 10.1161/JAHA.120.020364. Epub 2021 Aug 13. PMID 34387101
- [Derived] Shoamanesh A, Cassarly C, Morotti A, Romero JM, Oliveira-Filho J, Schlunk F, Jessel M, Butcher K, Gioia L, Ayres A, Vashkevich A, Schwab K, Afzal MR, Martin RH, Qureshi AI, Greenberg SM, Rosand J, Goldstein JN; ATACH-2 and NETT investigators. Intensive Blood Pressure Lowering and DWI Lesions in Intracerebral Hemorrhage: Exploratory Analysis of the ATACH-2 Randomized Trial. Neurocrit Care. 2022 Feb;36(1):71-81. doi: 10.1007/s12028-021-01254-9. Epub 2021 Jul 22. PMID 34292474
- [Derived] Fukuda-Doi M, Yamamoto H, Koga M, Doi Y, Qureshi AI, Yoshimura S, Miwa K, Ishigami A, Shiozawa M, Omae K, Ihara M, Toyoda K. Impact of Renal Impairment on Intensive Blood-Pressure-Lowering Therapy and Outcomes in Intracerebral Hemorrhage: Results From ATACH-2. Neurology. 2021 Aug 31;97(9):e913-e921. doi: 10.1212/WNL.0000000000012442. Epub 2021 Jul 1. PMID 34210824
- [Derived] Yogendrakumar V, Ramsay T, Menon BK, Qureshi AI, Saver JL, Dowlatshahi D. Hematoma Expansion Shift Analysis to Assess Acute Intracerebral Hemorrhage Treatments. Neurology. 2021 Aug 24;97(8):e755-e764. doi: 10.1212/WNL.0000000000012393. Epub 2021 Jun 18. PMID 34144995
- [Derived] Toyoda K, Palesch YY, Koga M, Foster L, Yamamoto H, Yoshimura S, Ihara M, Fukuda-Doi M, Okazaki S, Tanaka K, Miwa K, Hasegawa Y, Shiokawa Y, Iwama T, Kamiyama K, Hoshino H, Steiner T, Yoon BW, Wang Y, Hsu CY, Qureshi AI; ATACH-2 Trial Investigators. Regional Differences in the Response to Acute Blood Pressure Lowering After Cerebral Hemorrhage. Neurology. 2021 Feb 2;96(5):e740-e751. doi: 10.1212/WNL.0000000000011229. Epub 2020 Nov 20. PMID 33219136
- [Derived] Qureshi AI, Huang W, Lobanova I, Hanley DF, Hsu CY, Malhotra K, Steiner T, Suarez JI, Toyoda K, Yamamoto H; Antihypertensive Treatment of Cerebral Hemorrhage 2 Trial Investigators. Systolic Blood Pressure Reduction and Acute Kidney Injury in Intracerebral Hemorrhage. Stroke. 2020 Oct;51(10):3030-3038. doi: 10.1161/STROKEAHA.120.030272. Epub 2020 Aug 25. PMID 32838673
- [Derived] Fukuda-Doi M, Yamamoto H, Koga M, Palesch YY, Durkalski-Mauldin VL, Qureshi AI, Yoshimura S, Okazaki S, Miwa K, Okada Y, Ueda T, Okuda S, Nakahara J, Suzuki N, Toyoda K. Sex Differences in Blood Pressure-Lowering Therapy and Outcomes Following Intracerebral Hemorrhage: Results From ATACH-2. Stroke. 2020 Aug;51(8):2282-2286. doi: 10.1161/STROKEAHA.120.029770. Epub 2020 Jul 6. PMID 32623977
- [Derived] Qureshi AI, Foster LD, Lobanova I, Huang W, Suarez JI. Intensive Blood Pressure Lowering in Patients with Moderate to Severe Grade Acute Cerebral Hemorrhage: Post Hoc Analysis of Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH)-2 Trial. Cerebrovasc Dis. 2020;49(3):244-252. doi: 10.1159/000506358. Epub 2020 Jun 25. PMID 32585668
- [Derived] Toyoda K, Koga M, Yamamoto H, Foster L, Palesch YY, Wang Y, Sakai N, Hara T, Hsu CY, Itabashi R, Sato S, Fukuda-Doi M, Steiner T, Yoon BW, Hanley DF, Qureshi AI; ATACH-2 Trial Investigators. Clinical Outcomes Depending on Acute Blood Pressure After Cerebral Hemorrhage. Ann Neurol. 2019 Jan;85(1):105-113. doi: 10.1002/ana.25379. Epub 2019 Jan 7. PMID 30421455
- [Derived] Moullaali TJ, Wang X, Martin RH, Shipes VB, Qureshi AI, Anderson CS, Palesch YY. Statistical analysis plan for pooled individual patient data from two landmark randomized trials (INTERACT2 and ATACH-II) of intensive blood pressure lowering treatment in acute intracerebral hemorrhage. Int J Stroke. 2019 Apr;14(3):321-328. doi: 10.1177/1747493018813695. Epub 2018 Nov 12. PMID 30418098
- [Derived] Qureshi AI, Palesch YY, Foster LD, Barsan WG, Goldstein JN, Hanley DF, Hsu CY, Moy CS, Qureshi MH, Silbergleit R, Suarez JI, Toyoda K, Yamamoto H; ATACH 2 Trial Investigators. Blood Pressure-Attained Analysis of ATACH 2 Trial. Stroke. 2018 Jun;49(6):1412-1418. doi: 10.1161/STROKEAHA.117.019845. Epub 2018 May 22. PMID 29789395
- [Derived] Shoamanesh A, Morotti A, Romero JM, Oliveira-Filho J, Schlunk F, Jessel MJ, Ayres AM, Vashkevich A, Schwab K, Afzal MR, Cassarly C, Martin RH, Qureshi AI, Greenberg SM, Rosand J, Goldstein JN; Antihypertensive Treatment of Acute Cerebral Hemorrhage 2 (ATACH-2) and the Neurological Emergencies Treatment Trials (NETT) Network Investigators. Cerebral Microbleeds and the Effect of Intensive Blood Pressure Reduction on Hematoma Expansion and Functional Outcomes: A Secondary Analysis of the ATACH-2 Randomized Clinical Trial. JAMA Neurol. 2018 Jul 1;75(7):850-859. doi: 10.1001/jamaneurol.2018.0454. PMID 29710119
- [Derived] Morotti A, Boulouis G, Romero JM, Brouwers HB, Jessel MJ, Vashkevich A, Schwab K, Afzal MR, Cassarly C, Greenberg SM, Martin RH, Qureshi AI, Rosand J, Goldstein JN; ATACH-II and NETT investigators. Blood pressure reduction and noncontrast CT markers of intracerebral hemorrhage expansion. Neurology. 2017 Aug 8;89(6):548-554. doi: 10.1212/WNL.0000000000004210. Epub 2017 Jul 12. PMID 28701501
- [Derived] Morotti A, Brouwers HB, Romero JM, Jessel MJ, Vashkevich A, Schwab K, Afzal MR, Cassarly C, Greenberg SM, Martin RH, Qureshi AI, Rosand J, Goldstein JN; Antihypertensive Treatment of Acute Cerebral Hemorrhage II and Neurological Emergencies Treatment Trials Investigators. Intensive Blood Pressure Reduction and Spot Sign in Intracerebral Hemorrhage: A Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2017 Aug 1;74(8):950-960. doi: 10.1001/jamaneurol.2017.1014. PMID 28628707
- [Derived] Rodriguez-Luna D, Pineiro S, Rubiera M, Ribo M, Coscojuela P, Pagola J, Flores A, Muchada M, Ibarra B, Meler P, Sanjuan E, Hernandez-Guillamon M, Alvarez-Sabin J, Montaner J, Molina CA. Impact of blood pressure changes and course on hematoma growth in acute intracerebral hemorrhage. Eur J Neurol. 2013 Sep;20(9):1277-83. doi: 10.1111/ene.12180. Epub 2013 May 5. PMID 23647568
- [Derived] Toyoda K, Sato S, Koga M, Yamamoto H, Nakagawara J, Furui E, Shiokawa Y, Hasegawa Y, Okuda S, Sakai N, Kimura K, Okada Y, Yoshimura S, Hoshino H, Uesaka Y, Nakashima T, Itoh Y, Ueda T, Nishi T, Gotoh J, Nagatsuka K, Arihiro S, Yamaguchi T, Minematsu K. Run-up to participation in ATACH II in Japan. J Vasc Interv Neurol. 2012 Aug;5(supp):1-5. PMID 23230457
- [Derived] Sato S, Yamamoto H, Qureshi AI, Palesch YY, Toyoda K; ATACH-II study group. [Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH)-II at Japan site: study design and advance construction of domestic research network]. Rinsho Shinkeigaku. 2012;52(9):642-50. doi: 10.5692/clinicalneurol.52.642. Japanese. PMID 22989898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8,532 patients who presented to enrolling sites for emergency care within 6 hours of symptom onset and were found to have non-traumatic intracerebral hemorrhage (ICH) on head CT imaging were screened for eligibility beginning January 7, 2011. A total of 1000 patients were enrolled in the trial between May 15, 2011 and September 14, 2015.
Pre-assignment Details: Consent for participation was obtained from the patient or their allowable representative prior to randomization. All patients randomized were considered as enrolled. Treatment to lower systolic blood pressure (SBP) to the assigned range had to begin within 4.5 hours from symptom onset. Treatment for elevated SBP was not delayed for randomization.
Groups:
- Standard SBP Reduction Arm: Nicardipine hydrochloride was used according to need as the primary agent in lowering systolic blood pressure (SBP).
  The goal for the standard blood pressure reduction group was to reduce and maintain SBP under 180 mmHg for 24 hours from randomization. The target SBP for this treatment arm was approximately 160 mmHg (the center of the assigned treatment group range of SBP 140-179 mmHg).
  Nicardipine hydrochloride: IV nicardipine is initiated at a rate of 5 mg/hr, is continued, and is increased by 2.5 mg/hr increments every 15 min until the target SBP or maximum dose of 15 mg/hr is reached.
  If SBP was greater then the target SBP despite infusion of the maximum nicardipine dose for 30 minutes, a second agent could be used (Labetalol 5-20 mg IV bolus every 15 min; urapidil substituted in countries without labetalol available) for another hour. Nicardipine use was to be decreased incrementally or was discontinued if SBP fell below the assigned treatment range.
- Intensive SBP Reduction Arm: Nicardipine hydrochloride was used according to need as the primary agent in lowering systolic blood pressure (SBP).
  The goal for the intensive blood pressure reduction group was to reduce and maintain SBP under 140 mmHg for 24 hours from randomization. The target SBP for this treatment arm was 125 mmHg (the center of the treatment group range SBP 110 - 139 mmHg).
  Nicardipine hydrochloride: IV nicardipine is initiated at a rate of 5 mg/hr, is continued, and is increased by 2.5 mg/hr increments every 15 min until the target SBP or maximum dose of 15 mg/hr is reached.
  If SBP was greater than the target SBP after infusion of the maximum nicardipine dose for 30 min, a second agent could be used (Labetalol 5-20 mg IV bolus every 15 min; urapidil substituted in countries without labetalol available) for another hour. Nicardipine use was decreased incrementally or was discontinued if SBP fell below the assigned treatment range. Fluid bolus was given if needed for hypotension.
Period: Overall Study
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Started | 500 | 500
Completed | 480 | 481
Not Completed | 20 | 19
Not completed — Lost to Follow-up | 12 | 16
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Not Analyzed (any other reason) | 1 | 2

BASELINE CHARACTERISTICS:
Population: Subjects were randomized to standard vs. intensive SBP control. Below-range SBP was not artifically elevated in the standard SBP reduction arm; euvolemic fluid balance was maintained but spontaneous recovery was not prevented. For below-range SBP in the intensive SBP control arm, nicardipine was discontinued and if needed IV fluid bolus was given.
Groups:
- Standard SBP Reduction Arm: Nicardipine hydrochloride was used according to need as the primary agent in lowering systolic blood pressure (SBP).
  The goal for the standard blood pressure reduction group was to reduce and maintain SBP under 180 mmHg for 24 hours from randomization. The target SBP for this treatment arm was approximately 160 mmHg (the center of the assigned treatment group range of SBP 140-179 mmHg).
  Nicardipine hydrochloride: IV nicardipine is initiated at a rate of 5 mg/hr, is continued, and is increased by 2.5 mg/hr increments every 15 min until the target SBP or maximum dose of 15 mg/hr is reached.
  If SBP was greater than the target SBP despite infusion of the maximum nicardipine dose for 30 minutes, a second agent could be used (Labetalol 5-20 mg IV bolus every 15 min; urapidil substituted in countries without labetalol available) for another hour. Nicardipine use was to be decreased incrementally or was discontinued if SBP fell below the assigned treatment range.
- Total: Total of all reporting groups
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm | Total
Number analyzed (Participants) | 500 | 500 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (13.1) | 62 (13.1) | 61.93 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 196 | 380
  Male | 316 | 304 | 620
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity describes persons who have (versus have not) self-identified as being of Cuban, Mexican, Puerto Rican, Cuban, South or Central American, or other Spanish culture or origin, regardless of race.
  Data are analyzed according to the ethnicity and race of patients included to determine whether there are population differences in health measures or treatment responses that differ. Whether recruitment included an adequate diversity within the affected population is important to understanding the generalizability of results that were obtained and whether further research may be indicated.
  Participants
    Hispanic or Latino | 41 | 38 | 79
    Not Hispanic or Latino | 446 | 446 | 892
    Unknown or Not Reported | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnicity were recorded according to how a person identified themselves, not according to genetic testing or observation. The number of persons who reported American Indian, Alaska Native, Native Hawaiian of other Pacific Islander, or of having origins within more than one race has been included in the "other or unknown" category because the number of persons enrolled in the study from each of these categories was too small to provide a meaningful analysis that would examine these groups individually. Asian race included patients enrolled in Asian countries and non-Asian countries.
  Participants
    Race: Asian | 285 | 277 | 562
    Race: Black | 58 | 73 | 131
    Race: White | 145 | 142 | 287
    Race: Other or unknown | 12 | 8 | 20
Recruited at site in Asia [Count of Participants; unit: Participants] — Defined as patients who were enrolled at a clinical site geographically located within regions including Japan, China, Taiwan, or South Korea. Data from these patients were analyzed separately in addition to being part of the full group and other race/ethnicity analyses to examine for potential population differences surrounding intracerebral hemorrhage (ICH) events and recovery that are regional in nature.
  Participants | 273 | 264 | 537
First Glasgow Coma Scale Score assessed upon hospital emergency department (ED) arrival [Count of Participants; unit: Participants] — The Glasgow Coma Scale (GCS) score is a measure of level of consciousness. The scale quantifies response in three components: eye, motor, and verbal. A lower score indicates a reduced response and a higher score indicates a full response. At least one point is given in each category so the scale ranges from 3 to 15. A score of 3 indicates deep unconsciousness; a higher score indicates milder impairment of consciousness. The maximum score of 15 indicates consciousness is not impaired but other neurological symptoms may still be present. Estimated verbal scoring was used for intubated patients.
  Participants
    ED arrival GCS score = 3 - 11 | 74 | 73 | 147
    ED arrival GCS score = 12 - 14 | 142 | 152 | 294
    ED arrival GCS score = 15 | 284 | 275 | 559
Systolic Blood Pressure at presentation in hospital emergency department (ED) [Mean (Standard Deviation); unit: mmHg] — Blood pressure is reported as the systolic (systolic blood pressure or "SBP") reading "over" the diastolic (or DBP) reading, and is measured in millimeters of mercury (mmHg) on a gauge. SBP is a measure of the force pressing against the blood vessels when the heart contracts to push blood out to the body, and was considered most important for this study. DBP measures lingering pressure within the blood vessels as the heart fills with newly-oxygenated blood from the lungs. Hospitals selected the method that they felt was the most accurate way to report systolic blood pressures for each patient. Population: Data were missing for 1 patient in the standard-treatment group. It was permissible for pre-arrival or post-admission qualifying SBP to be used in eligibility determination if all other criteria were met.
  mmHg
    number analyzed (Participants) | 499 | 500 | 999
    (all) | 201.1 (26.9) | 200 (27.1) | 200.6 (27.0)
Median NIHSS score (range) [Median (Full Range); unit: units on a scale (NIHSS range 0 - 42)] — The National Institutes of Health Stroke Scale (NIHSS) is a serial measure of neurologic deficit (problems in function). It uses a scale (range 0 - 42) to quantify neurologic deficits in 11 categories. The categories are measured by asking questions that indicate the patient's level of consciousness, then testing horizontal eye movements, visual fields, facial palsy, movement in each limb, sensation, language and speech, and extinction or inattention on one side of the body. A score of 0 indicates normal function without neurologic deficit. Higher scores indicate greater severity of deficit.
  units on a scale (NIHSS range 0 - 42) | 11 [0 to 40] | 11 [0 to 40] | 11 [0 to 40]
Intracerebral Hematoma Volume [Median (Full Range); unit: cubic centimeters (cm3)] — Hematoma volumes are reported in cubic centimeters (cm3), as measured by the central reader. The area of the hematoma on head CT imaging was delineated by image analysis software with the use of density thresholds on each slice, followed by manual correction. The central reader and those performing manual correction were unaware of the patient identities, treatment assignments, clinical findings, and time points of image acquisition. The software provided total volume measurements by summing up volumes (product of area and slice thickness) from all the slices containing the hematoma. Population: A precise measure of bleeding within the brain was occasionally unable to be determined or baseline imaging wasn't submitted for analysis before data lock. This measure was missing for 8 patients in the standard treatment group and 4 in the intensive group. For eligibility, hematoma volume was estimated rapidly in 3 dimensions (ABC/2) at bedside.
  cubic centimeters (cm3)
    number analyzed (Participants) | 492 | 496 | 988
    (all) | 10.2 [0.98 to 79.1] | 10.3 [2.3 to 85.2] | 10.3 [0.98 to 85.2]
Intracerebral hematoma volume greater than 30 cm3 [Count of Participants; unit: Participants] — Hematoma volumes are reported in cubic centimeters (cm3), as measured by the central reader. The area of the hematoma on head CT imaging was delineated by image analysis software with the use of density thresholds on each slice, followed by manual correction. The central reader and those performing manual correction were unaware of the patient identities, treatment assignments, clinical findings, and time points of image acquisition. The software provided total volume measurements by summing up volumes (product of area and slice thickness) from all the slices containing the hematoma. Population: A precise measure of bleeding within the brain was occasionally unable to be determined or baseline imaging wasn't submitted for analysis before data lock. This measure was missing for 8 patients in the standard treatment group and 4 in the intensive group. For eligibility, hematoma volume was estimated rapidly in 3 dimensions (ABC/2) at bedside.
  Participants
    number analyzed (Participants) | 492 | 496 | 988
    (all) | 51 | 45 | 96
Intraventricular Hemorrhage [Count of Participants; unit: Participants] — Intraventricular hemorrhage is bleeding that is present within the ventricles, or internal fluid-filled spaces, within the brain. These spaces are usually filled with cerebrospinal fluid that also circulates around the brain and spinal column, which helps to protect and cushion the delicate brain tissue. In this study, when intraventricular hemorrhage was present it meant that bleeding had extended from another region within the brain tissue to also being present in the brain ventricles. Intraventricular blood is associated with other complications and may indicate a more severe condition. Population: The presence of blood within a brain ventricle as opposed to the hematoma (blood clot) within surrounding brain tissue pressing in to the ventricular space occasionally can't be determined, or baseline imaging wasn't submitted for analysis. This measure was missing for 8 patients in the standard treatment group and 4 in the intensive group.
  Participants
    number analyzed (Participants) | 492 | 496 | 988
    (all) | 142 | 122 | 264
Location of Hemorrhage [Count of Participants; unit: Participants] — The primary location of hemorrhage (bleeding) in the brain tissue was recorded as being located in the basal ganglia, thalamus, or a lobar region on either the right or left side of the brain. One patient was included that had a cerebellar hemorrhage, which means that bleeding was in the lower dorsal (back) region of the brain. Population: The primary location of bleeding within the brain is occasionally unable to be clearly determined, or baseline imaging wasn't submitted for analysis. This measure was missing for 8 patients in the standard treatment group and 4 in the intensive group.
  Participants
    number analyzed (Participants) | 492 | 496 | 988
    Thalamus | 180 | 193 | 373
    Basal ganglia | 251 | 255 | 506
    Cerebral lobe | 60 | 48 | 108
    Cerebellum | 1 | 0 | 1
Prior stroke/transient ischemic attack [Count of Participants; unit: Participants] | 84 | 80 | 164
Other prior nervous system disorders [Count of Participants; unit: Participants] | 17 | 23 | 40
History of congestive heart failure [Count of Participants; unit: Participants] | 21 | 16 | 37
History of atrial fibrillation [Count of Participants; unit: Participants] | 16 | 20 | 36
Myocardial infarction in the previous 3 months [Count of Participants; unit: Participants] | 0 | 1 | 1
History of coronary artery disease [Count of Participants; unit: Participants] | 17 | 27 | 44
History of hypertension [Count of Participants; unit: Participants] | 382 | 411 | 793
History of peripheral vascular disease [Count of Participants; unit: Participants] | 13 | 9 | 22
History of hyperlipidemia [Count of Participants; unit: Participants] | 119 | 122 | 241
History of cardiac dysrhythmias [Count of Participants; unit: Participants] | 21 | 17 | 38
History of diabetes mellitus Type 2 [Count of Participants; unit: Participants] | 83 | 92 | 175
Previous use of antihypertensive drugs [Count of Participants; unit: Participants] | 235 | 260 | 495
Symptom onset to randomization time, minutes [Mean (Standard Deviation); unit: minutes] | 184.7 (56.7) | 182.2 (57.2) | 183.5 (57)
Symptom onset to nicardipine infusion time [Mean (Standard Deviation); unit: minutes] — To qualify, patients had to have SBP greater than 180 mmHg prior to antihypertensive treatment and SBP not below 140 mmHg at the time of randomization. Nicardipine infusion had to be able to start within 4.5 hours of symptom onset. In accordance with recommendations, treatment of significant hypertension in patients presenting with ICH was not delayed for consent and randomization. This measure captures the earliest nicardipine start time but other intravenous antihypertensive medications may have been given before then. "Zero" nicardipine start rates may not have been recorded in all cases. Population: Data from 24 (3 intensive and 21 standard arm) patients was missing. If nicardipine wasn't needed to achieve the assigned SBP range at the time of randomization, more common in the standard arm, nicardipine was initiated at zero rate. "Zero rate" IV infusions have less consistent recording. Some patients had SBP within range without nicardipine.
  minutes
    number analyzed (Participants) | 479 | 497 | 976
    (all) | 165.3 (101.3) | 149 (65) | 157 (85.2)
Mean minimum systolic blood pressure, during the first 2 hours post randomization [Mean (Standard Deviation); unit: mmHg] — Population: Data were missing for 3 subjects in the standard treatment arm. If a vasoactive IV drip medication (such as nicardipine) is not in use, then standard-of-care parameters for close monitoring of SBP are different (frequency of required monitoring is less). Patient transfer and some procedures can preclude vigilance in recording research-only SBP.
  mmHg
    number analyzed (Participants) | 497 | 500 | 997
    (all) | 141.1 (14.8) | 128.9 (16) | 135 (16.6)
Failure to attain systolic blood pressure target within 2 hours [Count of Participants; unit: Participants] — Elevation of systolic blood pressure is common with intracerebral hemorrhage. Recovery of normalized blood pressure may occur quickly for some patients and only after an extended time for others, and more or less medication may be needed. The systolic blood pressure goal is usually achieved incrementally, as antihypertensive medication begins to take effect to control blood pressure. A lower target SBP range may take longer or be more difficult to achieve. The goal in this study was to achieve blood pressure control within 2 hours of randomization for all patients, regardless of treatment arm.
  Participants | 4 | 61 | 65
Failure to attain systolic blood pressure target for 2 consecutive hours during 2-24 hours [Count of Participants; unit: Participants] — This data parameter is a measure of the success (or lack of success) with which SBP control to the assigned treatment range was consistently maintained during the 24-hour SBP control study period.
  Participants | 7 | 78 | 85

OUTCOME MEASURES:

1. Primary Outcome: Death or Disability According to Modified Rankin Scale Score at 90 Days (3 Months) From Randomization
Description: The primary outcome was death or disability, defined by modified Rankin scale (mRS) of 4-6 at 90 days following treatment. The modified Rankin Scale score ranges from 0, indicating no symptoms, to 6, indicating death. A score of 4 indicates moderately severe disability including the inability to walk or attend to one's own bodily needs. A score of 5 indicates severe disability; bedridden, incontinent, and requiring constant nursing care. To score a 3 or lower on the mRS, a person must at least be able to walk without the assistance of another person. We chose the mRS because of its high inter-observer reliability, superiority to other indices, and consistency with previous trials in patients with ICH. Reliability was further increased by use of a structured interview template and by requiring mRS assessors to pass a certification test. Persons conducting the 90-day mRS assessment were to be unaware of the treatment arm or clinical course of the patients they assessed.
Time Frame: 90 days (± 14 days per protocol window; up to ± 30 days data is used) from randomization
Population: All subjects were analyzed for known death at any time following randomization. Patients surviving through 90 days (± 14 days per protocol window; data used up to ± 30 days) were assessed for disability using the mRS. Patients not completing the 90-day visit within 30 days of due date aren't included in the death & disability participant counts.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 500 | 500
Participants
  Death or disability at 90 days (mRS = 4 - 6) | 181 | 186
  Known death at or before 90 days | 34 | 33

2. Secondary Outcome: Quality of Life at 90 Days Using EuroQol (EQ) Measures: EQ-5D (EuroQol Five Dimension), Consisting of Standardized EQ-5D-3L (EuroQol Five Dimension, Three-Level) Questionnaire and EQ VAS (EuroQol Visual Analog Scale) Scores
Description: Standardized scales developed by the EuroQol Research Foundation were used as a secondary outcome measure in addition to the mRS scale score. The EQ-5D is a simple, standardized non-disease-specific instrument for describing and valuating health-related quality of life. The EQ-5D-3L questionnaire consists of 5 questions in 5 different domains and allows for responses from 1 (the best outcome) to 3 (the worst outcome) in each of five categories (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Total scores range from 5 to 15, with lower scores indicating better quality of life and a higher score indicating a worse quality of life. A second component of EuroQol outcome measurements is a printed 20 cm visual analogue scale (EQ VAS) that appears somewhat like a thermometer, on which a score from 0 (worst imaginable health state or death) to 100 (best imaginable health state) is marked by the patient (or, when necessary, their proxy) with the scale in view.
Time Frame: 90 days (± 14 days per protocol window; up to ± 30 days data is used) from randomization
Population: All available valid data were analyzed. Outcomes collected outside of 90 ± 30 days weren't considered valid. EQ-5D data were missing for 28 patients in the intensive group & for 27 in the standard group. EQ VAS data were missing for 144 patients in the intensive group and for 146 in the standard group.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 473 | 472
units on a scale
  EQ-5D utility scale questionnaire | 0.7 [0 to 1.0] | 0.7 [-0.109 to 1.0]
  EQ VAS (visual analog scale): number analyzed (Participants) | 354 | 356
  EQ VAS (visual analog scale) | 70 [0 to 100] | 62.5 [0 to 100]

3. Secondary Outcome: Hematoma Expansion (Number of Patients With Hematoma Expansion of 33% or Greater Between the Baseline and 24 +/- 6 Hours Head CTs, as Measured by the Central Reader for Patients With Readable Scans for Both Time Points Submitted by Data Lock.)
Description: Hematoma expansion as determined by serial CT scans: Hematoma expansion was defined as an increase in the volume of intraparenchymal hemorrhage of 33% or greater as measured by a central imaging analyst who was was unaware of the treatment assignments, clinical findings, and time points of image acquisition. The area of the hematoma was delineated by image analysis software with the use of density thresholds on each slice, followed by manual correction. To ensure accuracy and consistency of the readings, images were coded randomly and independently of subject numbers and manual correction was also done without awareness of treatment assignments, clinical findings, or time points of image acquisition. This data point is defined as being present (hematoma expansion of 33% or more was calculated between the baseline scan hematoma volume and the 24 +/- 6 hours hematoma volume measures at data analysis), meaning that hematoma expansion as defined must have occurred or it was not counted.
Time Frame: From the baseline head CT to the 24 +/- 6 hours from randomization head CT
Population: Participants with readable head CTs at baseline and 24 +/- 6 hours from randomization (submitted before data lock) were analyzed. Hematoma expansion was only recorded as present if ≥ 33% volume increase was calculated. Scans done outside of time window + margin, submitted after data lock, or not readable in standard DICOM format could not be used.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 426 | 450
Participants | 104 | 85

4. Other Pre Specified Outcome: Neurological Deterioration Within 24 Hours, Defined by a Decrease of 2 or More Points on the GCS Score or an Increase of 4 or More Points on the NIHSS Score From Baseline, Not Related to Sedation or Hypnotic-agent Use and Sustained for at Least 8 Hours.
Description: Neurologic deterioration was measured using two scales. The Glasgow Coma Scale (GCS) score measures of level of consciousness in eye, motor, and verbal components. At least one point is given in each category. The scale ranges from 3 to 15, with 3 indicating deep unconsciousness and 15 indicating consciousness is not impaired. The National Institutes of Health Stroke Scale (NIHSS) quantifies neurologic deficits in 11 categories. Level of consciousness, horizontal eye movement, visual fields, facial palsy, movement in each limb, sensation, language & speech, and extinction or inattention on one side of the body are tested. Scores range from 0 to 42, with 0 indicating normal function and higher scores indicating greater deficit severity. Neurological status was checked per ICU standards through 24 hours, recommended as hourly GCS and full assessment every 2 hours. NIHSS assessment at baseline and 24 +/- 3 hours was pre-specified. Assessments were added for suspected neurological change.
Time Frame: From randomization through the 24-hour treatment period
Population: All subjects were assessed for neurological status regularly. Grid-estimated verbal scoring based on eye and motor scores was used for intubated patients so that GCS scores could be compared over time and was consistent across patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 500 | 500
Participants | 40 | 55

5. Other Pre Specified Outcome: Hypotension Within 72 Hours
Description: Hypotension (abnormally low blood pressure) was the most likely adverse event that could be associated with the study treatment, and is the primary basis (risk) on which neurological deterioration or other untoward effects of the study treatment could occur. It is therefore examined as a numerically-measured occurrence in addition to monitoring patients closely for neurological deterioration or other symptoms. Hypotension, when named as an adverse event, was defined as the syndrome of low blood pressure with SBP < 85 mmHg. Instances of hypotension were to be avoided through close monitoring, and administration of fluid bolus for SBP < 110 mmHg. If hypotension did occur, it was to be reversed as quickly as possible through discontinuation of intravenous nicardipine and intravenous fluid administration, which can be accomplished readily in a variety of settings where patients with intracerebral hemorrhage are routinely housed during early hospitalization.
Time Frame: From randomization through 72 hours from randomization
Population: Blood pressure including the potential for hypotension was monitored according to intensive care unit standards for ICH patients during early hospitalization. Blood pressure was monitored more closely during the 24-hour study period and at times when nicardipine (or other/secondary IV antihypertensive medications) were being titrated.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 500 | 500
Participants | 3 | 6

6. Other Pre Specified Outcome: Treatment-related Serious Adverse Event Within 72 Hours of Randomization
Description: Adverse events (AEs) and serious adverse events (SAEs) were assessed by the site investigators for all patients, including for their potential relatedness to the study treatment. An Independent Oversight Committee (IOC) reviewed and adjudicated all adverse event data. The 72-hours-from-randomization time window was considered the most likely time frame during which treatment-related adverse events or serious adverse events would be observed. Terminology from the Medical Dictionary for Regulatory Activities (MedDRA) and severity criteria from the Common Terminology Criteria for Adverse Events (CTCAE v. 4.03) were used as a basis for reporting adverse events. Serious adverse events are defined as being fatal, life-threatening, resulting in hospitalization or prolonged hospitalization, resulting in disability or congenital anomaly, or requiring intervention to prevent permanent impairment or damage and were required to be reported promptly.
Time Frame: From randomization through 72 hours (3 days)
Population: Relatedness is defined by the terms unrelated, unlikely, possibly, probably, or definitely related to the study treatment. Results are entered as the count of participants experiencing any serious adverse event within 72 hours of randomization that was determined by the site investigator to possibly or more have relationship to the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 500 | 500
Participants | 6 | 8

7. Other Pre Specified Outcome: Any Serious Adverse Event Within the 90-day Study Period
Description: The complete count of all subjects who experienced any serious adverse events throughout their participation in the trial was included in this tabulation. Adverse events (AEs) and serious adverse events (SAEs) were assessed by the site investigators for all patients. Potential relatedness to the study treatment was a required reporting element for all adverse events but was not considered in this count. Terminology from the Medical Dictionary for Regulatory Activities (MedDRA) and severity criteria from the Common Terminology Criteria for Adverse Events (CTCAE v. 4.03) were used as a basis for reporting adverse events. Serious adverse events are defined as being fatal, life-threatening, resulting in hospitalization or prolonged hospitalization, resulting in disability or congenital anomaly, or requiring intervention to prevent permanent impairment or damage and were required to be reported promptly. An Independent Oversight Committee (IOC) reviewed and adjudicated adverse event data.
Time Frame: From randomization through the 90 day visit (90 ± 14 days per protocol window; up to ± 30 days data is used) or until known death, withdrawal, or loss to follow-up.
Population: Patients may have experienced more than one adverse event. This measure is designed to show the total count of any patients who experienced any type of serious adverse event, whether it was felt to be related to the study treatment or not, throughout the duration of their participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Number analyzed (Participants) | 500 | 500
Participants | 100 | 128

ADVERSE EVENTS:
Time Frame: Adverse events were collected between randomization and the end-of-study visit. All adverse events (defined as abnormal test results, new diagnoses, worsening of conditions, or other health events of clinical significance) were collected through day 7 or hospital discharge, whichever came first. Only serious adverse events (SAEs) were collected from Day 7 (or discharge, if sooner) through final study visits at 3-months +/- 30 days. SAEs, 5-day reporting timeline.
Description: Adverse events during hospitalization: assessed from medical records. Post-hospital discharge, patients/proxy were asked if illness or hospitalization had occurred; available medical records also checked. CTCAE v. 4.03 as severity grading reference. Relatedness of adverse events: assessed by the site investigator within categories unrelated, unlikely, possibly, probably, or definitely related to the study treatment. Analyses by code + related safety groupings. AEs ≩ all subjects being affected.
Arm/Group | Standard SBP Reduction Arm | Intensive SBP Reduction Arm
Serious Adverse Events (participants affected / at risk) | 100/500 | 128/500
Other Adverse Events (participants affected / at risk) | 500/500 | 500/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard SBP Reduction Arm (N=500) | Intensive SBP Reduction Arm (N=500)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angiopathy (Cardiac disorders) | 0 (0) | 1 (1) — Coded under vascular disorders, also analyzed with cardiac disorders for safety
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blood creatinine increased (Renal and urinary disorders) | 1 (1) | 0 (0) — Coded under investigations, also analyzed with renal disorders for safety
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Brain herniation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Brain oedema (Nervous system disorders) | 2 (2) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CNS ventriculitis (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 4 (4)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 6 (6) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Cerebrovascular accident (Nervous system disorders) | 19 (19) | 17 (17)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0) — (Meeting SAE criteria); coded under general disorders, also analyzed with cardiac disorders for safety
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2) — (Meeting SAE criteria)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Circulatory collapse (Vascular disorders) | 0 (0) | 2 (2)
Clostridial infection (Infections and infestations) | 1 (1) | 1 (1) — (Meeting SAE criteria)
Convulsion (Nervous system disorders) | 3 (3) | 1 (1) — (Meeting SAE criteria)
Cranioplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Cyst aspiration (Investigations) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 3 (3) — (Meeting SAE criteria)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2) — (Meeting SAE criteria)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) — (Meeting SAE criteria)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Haemorrhage (Vascular disorders) | 2 (2) | 1 (1) — (Meeting SAE criteria)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 3 (3) — (Meeting SAE criteria)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Haemorrhagic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Hydrocephalus (Nervous system disorders) | 4 (4) | 7 (7) — (Meeting SAE criteria)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Hypertension (Cardiac disorders) | 1 (1) | 3 (3) — (Meeting SAE criteria); coded under general disorders, also analyzed with cardiac disorders for safety
Hypertensive crisis (Cardiac disorders) | 0 (0) | 1 (1) — Coded under vascular disorders, also analyzed with cardiac disorders for safety
Hypertensive emergency (Cardiac disorders) | 0 (0) | 1 (1) — Coded under vascular disorders, also analyzed with cardiac disorders for safety
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — (Meeting SAE criteria)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) — (Meeting SAE criteria); coded under vascular disorders, also analyzed with cardiac disorders for safety
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (2) — (Meeting SAE criteria)
Ischaemia (Nervous system disorders) | 1 (1) | 0 (0) — Coded under vascular disorders, also analyzed with brain infarct/nervous disorders for safety
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) — (Meeting SAE criteria)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Mental impairment (Nervous system disorders) | 1 (1) | 2 (2) — (Meeting SAE criteria)
Mental status changes (Nervous system disorders) | 2 (2) | 0 (0) — (Meeting SAE criteria)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 9 (9) | 18 (18) — (Meeting SAE criteria)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 1 (1) — (Meeting SAE criteria)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Pneumonia (Infections and infestations) | 5 (5) | 9 (9) — (Meeting SAE criteria)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (9) — (Meeting SAE criteria)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) — (Meeting SAE criteria)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) — (Meeting SAE criteria)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 4 (4) — (Meeting SAE criteria)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — (Meeting SAE criteria)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (10) — (Meeting SAE criteria)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1)
Schizophrenia, paranoid type (Psychiatric disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) — (Meeting SAE criteria)
Stroke in evolution (Nervous system disorders) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — (Meeting SAE criteria)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — (Meeting SAE criteria)
Urosepsis (Infections and infestations) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard SBP Reduction Arm (N=500) | Intensive SBP Reduction Arm (N=500)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — (AE Not meeting SAE criteria)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Administration site reaction (General disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 6 (7) | 13 (14)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 9 (9)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Aortic stenosis (Cardiac disorders) | 0 (0) | 1 (1) — Coded under vascular disorders, also analyzed with cardiac disorders for safety
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) — (AE Not meeting SAE criteria)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — (AE Not meeting SAE criteria)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 6 (7) — (AE Not meeting SAE criteria)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — (AE Not meeting SAE criteria)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Blood chloride abnormal (Investigations) | 0 (0) | 1 (1)
Blood chloride increased (Investigations) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine abnormal (Renal and urinary disorders) | 1 (1) | 0 (0) — Coded under investigations, also analyzed with renal disorders for safety
Blood creatinine decreased (Renal and urinary disorders) | 0 (0) | 1 (1) — Coded under investigations, also analyzed with renal disorders for safety
Blood creatinine increased (Renal and urinary disorders) | 2 (2) | 6 (6) — (AE Not meeting SAE criteria) Coded under investigations, also analyzed with renal disorders for safety.
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Blood pressure decreased (Cardiac disorders) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Cardiac disorders) | 1 (1) | 0 (0) — Coded under investigations, also analyzed with cardiac disorders for safety
Blood pressure increased (Cardiac disorders) | 1 (1) | 0 (0) — Coded under investigations, also analyzed with cardiac disorders for safety
Blood sodium increased (Investigations) | 0 (0) | 1 (1)
Blood urea decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood urea increased (Renal and urinary disorders) | 3 (3) | 2 (2)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 5 (5) | 1 (1) — (AE Not meeting SAE criteria)
Brain oedema (Nervous system disorders) | 1 (1) | 5 (5) — (AE Not meeting SAE criteria)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) — (AE Not meeting SAE criteria)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Cardiac murmur (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 6 (6)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 1 (1) — (AE Not meeting SAE criteria)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2) — (AE Not meeting SAE criteria)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (5) | 4 (5) — (AE Not meeting SAE criteria)
Chest discomfort (Cardiac disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 2 (2) | 3 (3) — (AE Not meeting SAE criteria); coded under general disorders, also analyzed with cardiac disorders for safety
Chills (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — (AE Not meeting SAE criteria)
Clostridial infection (Infections and infestations) | 3 (3) | 0 (0) — (AE Not meeting SAE criteria)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Coma scale abnormal (Investigations) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Consciousness fluctuating (Nervous system disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (25) | 25 (25)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 7 (7) | 4 (4) — (AE Not meeting SAE criteria)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Craniotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 1 (1) — (AE Not meeting SAE criteria)
Delirium (Psychiatric disorders) | 7 (7) | 8 (8)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1) — (AE Not meeting SAE criteria)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) — (AE Not meeting SAE criteria)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (6)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — (AE Not meeting SAE criteria)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) — (AE Not meeting SAE criteria)
Dysuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Electrocardiogram ST segment depression (Cardiac disorders) | 1 (1) | 0 (0) — Coded under investigations, also analyzed with cardiac disorders for safety
Electrolyte imbalance (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Endotracheal intubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) — (AE Not meeting SAE criteria)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 5 (5) — (AE Not meeting SAE criteria)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fluid overload (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastric occult blood positive (Investigations) | 0 (0) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Glomerular filtration rate increased (Renal and urinary disorders) | 0 (0) | 1 (1) — Coded under investigations, also analyzed with renal disorders for safety
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) — (AE Not meeting SAE criteria)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) — (AE Not meeting SAE criteria)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 8 (9) — (AE Not meeting SAE criteria)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Hallucination (Psychiatric disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 22 (25) | 17 (18)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (4) | 3 (3) — (AE Not meeting SAE criteria)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 4 (4) | 5 (5) — (AE Not meeting SAE criteria)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) — (AE Not meeting SAE criteria)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 11 (11) | 10 (10)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (3)
Hypertension (Cardiac disorders) | 5 (6) | 3 (3) — (AE Not meeting SAE criteria); coded under vascular disorders, also analyzed with cardiac disorders for safety
Hypervolaemia (Renal and urinary disorders) | 0 (0) | 1 (1) — Coded under metabolism and nutrition disorders, also analyzed with renal disorders for safety
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) — (AE Not meeting SAE criteria)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (32) | 38 (39)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (16) | 6 (6) — (AE Not meeting SAE criteria)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (8) | 9 (9)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 3 (3) | 6 (6) — (AE Not meeting SAE criteria); coded under vascular disorders, also analyzed with cardiac disorders for safety
Hypovolaemia (Renal and urinary disorders) | 0 (0) | 1 (1) — Coded under metabolism and nutrition disorders, also analyzed with renal disorders for safety
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — (AE Not meeting SAE criteria)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 3 (3) | 3 (3)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 0 (0) — (AE Not meeting SAE criteria)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 3 (3)
Laboratory test abnormal (Investigations) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 12 (12) — (AE Not meeting SAE criteria)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 4 (4)
Liver function test abnormal (Investigations) | 2 (3) | 2 (2) — (AE Not meeting SAE criteria)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 12 (14) | 14 (14) — (AE Not meeting SAE criteria)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (2) — (AE Not meeting SAE criteria)
Mental impairment (Nervous system disorders) | 1 (1) | 2 (2) — (AE Not meeting SAE criteria)
Mental status changes (Nervous system disorders) | 4 (4) | 2 (2) — (AE Not meeting SAE criteria)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 8 (8)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 3 (3) | 8 (8) — (AE Not meeting SAE criteria)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (2) — (AE Not meeting SAE criteria)
PO2 decreased (Investigations) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Partial seizures (Nervous system disorders) | 3 (4) | 0 (0) — (AE Not meeting SAE criteria)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 18 (18) | 17 (17)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Pneumocephalus (Nervous system disorders) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 11 (12) | 18 (20) — (AE Not meeting SAE criteria)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 21 (23) — (AE Not meeting SAE criteria)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post transfusion purpura (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — (AE Not meeting SAE criteria)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 39 (40) | 30 (32) — (AE Not meeting SAE criteria)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) — (AE Not meeting SAE criteria)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 13 (13) — (AE Not meeting SAE criteria)
Renal function test abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 3 (3) | 6 (6)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — (AE Not meeting SAE criteria)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — (AE Not meeting SAE criteria)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (2) | 2 (2)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scleral oedema (Eye disorders) | 1 (1) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (2) | 4 (4)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) — (AE Not meeting SAE criteria)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Sputum culture positive (Investigations) | 1 (1) | 0 (0)
Sputum increased (Investigations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Stereotactic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0)
Stress ulcer (Gastrointestinal disorders) | 3 (3) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — (AE Not meeting SAE criteria)
Tachycardia (Cardiac disorders) | 7 (7) | 8 (9) — (AE Not meeting SAE criteria)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Troponin I increased (Cardiac disorders) | 2 (3) | 1 (1)
Troponin increased (Cardiac disorders) | 3 (3) | 6 (7)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1) — (AE Not meeting SAE criteria)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 24 (24) | 20 (20) — (AE Not meeting SAE criteria)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Urine output decreased (Renal and urinary disorders) | 0 (0) | 6 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (11) | 13 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 3 (3) | 4 (4)

LIMITATIONS AND CAVEATS:
Treatment failures, randomization window, demographics, pre-randomization treatment, low death/disability, favorable baselines, and early termination could limit generalizability of primary (all with intent-to-treat) results and some sub-analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The overall Principal Investigator IS, but the Data Coordination Unit (statistical) Principal Investigator IS NOT employed by the sponsor. Prior to release of a public-use data set, any study PIs/other collaborators may submit a proposal requesting data access, assistance with statistical analyses, and publication of additional results. All proposals are reviewed by a Publications Committee that includes the primary study PI, the statistical PI, the NINDS project scientist, and appointed others.